CLINICAL TRIAL: NCT01992601
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Investigate the Pharmacokinetic Drug Interaction Between Rosuvastatin and Telmisartan in Healthy Volunteer
Acronym: YH16410 DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: YH16410-101
Record Dates: First submitted 2013-09-30; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Healthy Volunteer
Keywords: Drug interaction; Rosuvastatin; Telmisartan; Pharmacokinetic; (Pharmacokinetics and Drug Interaction)
MeSH Terms: interventions — Rosuvastatin Calcium; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): This arm is consist of 12 subject. Crestor 20mg alone for 6 day during period 1. Crestor 20mg and Micardis 80mg for 6 day during period 2.
  Interventions: Drug: Crestor 20mg(Rosuvastatin 20mg), Micardis 80mg(Telmisartan 80mg)
- 2 (Experimental): This arm is consist of 12 subject. Crestor 20mg and Micardis 80mg for 6 day during period 1. Crestor 20mg alone for 6 day during period 2.
  Interventions: Drug: Crestor 20mg(Rosuvastatin 20mg), Micardis 80mg(Telmisartan 80mg)
- 3 (Experimental): This arm is consist of 12 subject. Micardis 80mg alone for 6 day during period 1. Crestor 20mg and Micardis 80mg for 6 day during period 2.
  Interventions: Drug: Crestor 20mg(Rosuvastatin 20mg), Micardis 80mg(Telmisartan 80mg)
- 4 (Experimental): This arm is consist of 12 subject. Crestor 20mg and Micardis 80mg for 6 day during period 1. Micardis 80mg alone for 6 day during period 2.
  Interventions: Drug: Crestor 20mg(Rosuvastatin 20mg), Micardis 80mg(Telmisartan 80mg)

INTERVENTIONS:
Drug: Crestor 20mg(Rosuvastatin 20mg), Micardis 80mg(Telmisartan 80mg) — For co-administration, Crestor 1 tablet and Micardis 1 tablet a day for 6 days in each period.
  For separate administration, Crestor 1 tablet a day for 6 days and Micardis 1 tablet a day for 6 days in each period.

SUMMARY:
This clinical trial is designed to compare the pharmacokinetic characteristics of combination and separate administration of Crestor(Rosuvastatin) and Micardis(Telmisartan). Also investigate drug interaction between separate and combination administration.

Total number of subjects is 48. 4 group(12 for 1 group), 2 period, consecutive 6 day administration, 16 days washout after 6th day of administration.

The subjects of Part 1 take Crestor alone and Crestor+Micardis combination by a cross-over design during 2 each period.

The other subjects of Part 2 take Micardis alone and Crestor+Micardis combination by a cross-over design during 2 each period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female aged 20 to 50 with a body mass index(BMI) between 19 and 27 kg/m2
2. Acceptable medical history, physical examination, laboratory tests and EKG, during screening
3. Provision of signed written informed consent •20~50 yrs old, healthy Korean Subjects

Exclusion Criteria:

1.History of and clinically significant disease 2.Sitting blood pressure meeting the following criteria at screening: 150 ≤ systolic blood pressure ≤90 (mmHg) and 95 ≤ diastolic blood pressure ≤ 50 (mmHg) amd 100 ≤ Heart rate ≤ 40 3. A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs.

4. Administration of other investigational products within 90 days prior to the first dosing.

5. Administration of herbal medicine within 30 days or administration of ethical drugs within 14 days or administration of over-the-counter (OTC) drugs within 7 days prior to the first dosing of the investigational product (if the investigator (study doctor) determines that the person meets other criteria appropriately, the relevant person may participate in the study).

6.Have AST(SGOT) or/and ALT(SGPT) > 3 times of normal upper limit at the time of screening 7. Volunteers considered not eligible for the clinical trial by the investigator (study doctor) due to reasons including laboratory test results, ECGs, or vital signs.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
AUC | 72hr
  AUC τ,ss of Rosuvastatin and Telmisartan
Cmax | 72hr
  Cmax,ss of Rosuvastatin and Telmisartan

SECONDARY OUTCOMES:
AUC | 72hr
  AUC last,ss of Rosuvastatin, N-desmetyl Rosuvastatin and Telmisartan
AUC | 72hr
  AUC inf,ss of Rosuvastatin, N-desmetyl Rosuvastatin and Telmisartan
Tmax | 72hr
  Tmax,ss of Rosuvastatin, N-desmetyl Rosuvastatin and Telmisartan
t1/2 | 72hr
  t1/2 of Rosuvastatin, N-desmetyl Rosuvastatin and Telmisartan
Cmin | 72hr
  Cmin,ss of Rosuvastatin, N-desmetyl Rosuvastatin and Telmisartan
AUC | 72hr
  AUCτ,ss of N-desmetyl Rosuvastatin
Cmax | 72hr
  Cmax,ss of N-desmetyl Rosuvastatin

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University, Seoul, South Korea

REFERENCES:
- [Derived] Son M, Kim Y, Lee D, Roh H, Son H, Guk J, Jang SB, Nam SY, Park K. Pharmacokinetic interaction between rosuvastatin and telmisartan in healthy Korean male volunteers: a randomized, open-label, two-period, crossover, multiple-dose study. Clin Ther. 2014 Aug 1;36(8):1147-58. doi: 10.1016/j.clinthera.2014.06.007. Epub 2014 Jul 3. PMID 24998012